CLINICAL TRIAL: NCT01751659
Title: Clinician Attitudes and Behaviors Regarding Use of Pre-Exposure Prophylaxis (PrEP) for Primary HIV Prevention
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: ATN 111
Record Dates: First submitted 2012-12-14; First posted 2012-12-18 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2016-11

CONDITIONS: Clinician Attitudes About PrEP

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Phase I: * Semi-structured face-to-face or telephone interviews of 10 ATN-affiliated clinicians.
  * The total duration of Phase 1 is expected to last approximately nine months, including data analysis.
- Phase II: * Development of a new theory-based survey instrument and cognitive interview testing of this survey with approximately five clinicians (of those who participated in Phase 1).
  * The total duration of Phase 2 is expected to last approximately three months, including qualitative analysis of the interviews and modification of the survey.
- Phase III: * Administration of the newly developed survey to approximately 60 ATN-affiliated clinicians.
  * The total duration of Phase 3 will last approximately six to nine months.

SUMMARY:
This is a three phase study designed to examine clinician behaviors with regard to recommending and prescribing pre-exposure prophylaxis (PrEP) as a primary Human Immunodeficiency Virus (HIV) prevention strategy, and to identify knowledge-related and attitudinal factors associated with these behaviors. Each phase consists of the following:

Phase 1: Semi-structured face-to-face or telephone interviews of ATN-affiliated clinicians. Approximately 10 clinicians will be interviewed.

Phase 2: Development of a new theory-based survey instrument and cognitive interview testing of this survey. Approximately five clinicians (of those who participated in Phase 1) will be interviewed.

Phase 3: Administration of the newly developed survey to ATN-affiliated clinicians. Approximately 60 clinicians will be interviewed.

ELIGIBILITY:
Inclusion Criteria:

* Clinicians (including physicians, nurse practitioners, and physician assistants) that EITHER: Provide primary HIV care for HIV-infected and primary care for HIV-uninfected adolescents; OR Provide primary HIV care to HIV-infected adolescents only;
* Provides services to adolescents and young adults at ATN sites or one of their community partners;
* Ability to understand spoken English; and
* For Phase 2 only: prior participation in Phase 1.

Exclusion Criteria:

* Intoxicated or under the influence of alcohol or other substances at the time of consent;
* Visibly distraught and/or visibly emotionally unstable (i.e., exhibiting suicidal, homicidal, or violent behavior) and in the opinion of the protocol chair would interfere with the ability to give true informed consent; and
* For Phase 3 only: prior participation in Phase 1 or 2 of this study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: ATN-affiliated clinicians (including physicians, nurse practitioners, and physician assistants) who EITHER 1) provide care for HIV-infected and HIV-uninfected adolescents OR 2) provide care to HIV-infected adolescents only.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2012-09; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Explore clinician attitudes and prescribing behaviors in MSM and heterosexually active adults | 2 years
  Explore clinician attitudes and prescribing behaviors with regard to the use of PrEP in men who have sex with men (MSM) and heterosexually active adults as described in the current CDC guidelines, as well as in MSM and heterosexually active adolescents, who are not specifically covered by the guidelines
Identify factors associated with prescribing PrEP | 2 years
  Identify factors associated with prescribing PrEP, in a sample of clinicians who provide care to HIV-infected adolescents alone OR to HIV-infected and HIV-uninfected adolescents.

SECONDARY OUTCOMES:
Explore clinician attitudes toward the use of PrEP in potential target populations other than MSM and heterosexually active adults. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Mullins, MD, Study Chair — Adolescent Trials Network
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- See also: ATN website — http://www.atnonline.org